CLINICAL TRIAL: NCT05183555
Title: Early Feasibility Study of Somatostatin Receptors PET Imaging (68Ga-DOTATOC PET/CT) for the Diagnosis of Infective Endocarditis
Brief Title: Early Feasibility Study of Somatostatin Receptors PET Imaging for the Diagnosis of Infective Endocarditis
Acronym: DOTENDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021PI119
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Intervention Model Description: Single-center, early feasibility clinical trial (RIPH1 type) using a radiopharmaceutical (drug) off-label.
  This study is based on the evaluation of an off-label radiopharmaceutical, 68Ga-DOTATOC in PET/CT, to detect infective endocarditis. The marketing authorization of 68Ga-DOTATOC is for the neuroendocrine tumors assessment (NET). Currently, a clinical study using 68Ga-DOTATOC PET/CT to detect myocarditis in the inflammatory phase is conducted by a team of the CHRU of Nancy Fourteen patients with definite IE according to the modified Duke criteria (Li) will be included and referred for 18F-FDG PET/CT in the study. A 68Ga-DOTATOC PET/CT scan will be performed specifically for research at 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with definite IE will be included and referred for 18F-FDG PET/CT in the study (Experimental): Fourteen patients with definite IE according to the modified Duke criteria (Li) will be included and referred for 18F-FDG PET/CT in the study. A 68Ga-DOTATOC PET/CT scan will be performed specifically for research at 24 hours.
  Interventions: Drug: 68Ga-DOTATOC PET/CT

INTERVENTIONS:
Drug: 68Ga-DOTATOC PET/CT — 68Ga-DOTATOC PET/CT will be recorded the following day of 18F-FDG PET/CT if patient signed the consent
  Other Names: 18F-FDG PET/CT

SUMMARY:
Study hypothesis: 68Ga-DOTATOC PET/CT could detect cardiac foci of infective endocarditis regardless of the type of valve (native or prosthetic) and also extracardiac localizations related to this pathology (infection responsible, peripheral emboli, ...). This study is a proof of concept with low population

DETAILED DESCRIPTION:
The incidence of infective endocarditis (IE) in France is estimated to be around 30 cases per million inhabitants in studies conducted in Western countries and is significantly increased in patients with a valve prosthesis and even more so in cases of a history of endocarditis. The morbi-mortality is significant and the hospital mortality rate is 20%.

The diagnosis of IE remains difficult and according to the modified Duke criteria, the diagnostic sensitivity is 80%.

Currently, the diagnosis of IE is often determined according to the 2015 ESC criteria and the sensitivity increases from 57% to 84% regarding IE on prosthetic valves.

The 18F-FDG PET/CT examination is of major interest in the diagnosis of AR on prosthetic valves with a detection sensitivity of between 70 and 90% (with an accuracy of 70 to 80%). Concerning native valves, the sensitivity of PET/CT remains below 50%.

Indeed, a "physiological" myocardial fixation in 18F-FDG PET/CT compromises the interpretation of PET exam, so it is important to start a hypoglycemic-hyperlipidic diet the day before the 18F-FDG PET/CT, followed by a 12-hour fasting period.

For several years, a radiopharmaceutical, 68Ga-DOTATOC (68Ga-edotreotide) has been used in PET/CT for the diagnosis and follow-up of neuroendocrine tumours (NETs). 68Ga-DOTATOC binds mainly with high affinity to somatostatin receptor subtype 2 (SSTR2) but also to somatostatin receptor subtype 5 (SSTR5).

Activated monocytes, macrophages, and lymphocytes express somatostatin receptors , thus detection of SSTR2 receptors expressed by inflammatory cells could help for the diagnosis of infective endocarditis.

PET/CT with 68Ga-DOTATOC could thus detect inflammatory cells at infectious sites. This radiopharmaceutical has already shown an ability to identify a myocardial inflammation (inflammatory phase myocarditis and cardiac sarcoidosis).

In current study conducted by our teams (NCT03347760 on ClinicalTrials.gov), early results showed the capacity of the 68Ga-DOTATOC to detect efficiently myocarditis, including myocarditis induced by RNA anti-COVID vaccinations.

In vitro, the 18FDG uptake by inflammatory cells is more important than the 68Ga-DOTATOC uptake, but the contrast between infection focus and healthy tissue should be better since 68Ga-DOTATOC does not cause any physiological myocardial uptake. The 68Ga-DOTATOC does not required any special metabolic preparation or prolonged fasting often poorly supported by patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult who has received full information about the organisation of the research and has signed informed consent adult
* Participant hospitalised for definite AE according to modified Duke criteria (Li), on native or prosthetic valve, referred for 18F-FDG PET/CT from Cardiology and Infectious Diseases departments

Exclusion Criteria:

* Person with a history of hypersensitivity from previous use of 68Ga-DOTATOC
* Unable to perform a 68Ga-DOTATOC PET scan (agitated, confused patient...).
* Inability to schedule 68Ga-DOTATOC PET/CT the day after 18F-FDG PET/CT.
* Person with severe renal impairment (GFR <30 ml/min/1.73 m2)
* Participant treated with a somatostatin analogue.
* Participant with Cushing's syndrome
* Pregnant, potentially pregnant or breastfeeding women
* Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person of full age who is unable to give consent
* Person deprived of liberty by a judicial or administrative decision
* Person subject to psychiatric care by virtue of Articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Detectability of infective endocarditis by 68Ga-DOTATOC PET/CT | one year
  to visually evaluate the detectability of cardiac and extracardiac foci associated with infective endocarditis (IE) on native or prosthetic valve by 68Ga-DOTATOC PET/CT.

SECONDARY OUTCOMES:
To quantify the infective foci uptake of 68Ga-DOTATOC | one year
  To quantify the infective foci uptake of 68Ga-DOTATOC with measure of Standard Uptake Value (SUV) related to blood activity.
68Ga-DOTATOC PET/CT and 18F-FDG PET/CT results comparison | one year
  To compare 68Ga-DOTATOC PET/CT results with 18F-FDG PET/CT results, of visual and quantitative analysis on whole body PET/CT
68Ga-DOTATOC PET/CT and 18F-FDG PET/CT results comparison of cardiac step | one year
  3. To compare the 68Ga-DOTATOC PET/CT results with those of 18F-FDG PET/CT, of visual and quantitative analysis of cardiac step recordings

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No